CLINICAL TRIAL: NCT02195180
Title: Phase II, Randomized, Controlled, Clinical Trial Exploring Efficacy and Safety of ERY001 (L-asparaginase Encapsulated in Red Blood Cells) in Association With Gemcitabine or FOLFOX4 in Second-line Therapy for Patients With Progressive Metastatic Pancreatic Carcinoma
Brief Title: Efficacy and Safety of L-asparaginase Encapsulated in RBC Combined With Gemcitabine or FOLFOX in 2nd Line for Progressive Metastatic Pancreatic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ERYtech Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRASPANC 2013-03; 2013-004262-34 (EudraCT Number)
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2017-11

CONDITIONS: Pancreatic Adenocarcinoma Metastatic
Keywords: Pancreas; adenocarcinoma; cancer; asparaginase; erythrocytes; red blood cell; Encapsulation; folfox; gemcitabine
MeSH Terms: conditions — Adenocarcinoma; Neoplasms | interventions — Erythrocyte Count; Gemcitabine; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard of care combined with ERY001 (Experimental): standard of care = Gemcitabine or folfox
  Interventions: Drug: ERY001; Drug: Gemcitabine; Drug: 5-fluoro-uracil/oxaliplatin/leucovorin (folfox)
- standard of care alone (Sham Comparator): standard of care = Gemcitabine or folfox
  Interventions: Drug: Gemcitabine; Drug: 5-fluoro-uracil/oxaliplatin/leucovorin (folfox)

INTERVENTIONS:
Drug: ERY001
  Other Names: L asparaginase encapsulated in erythrocytes
  Arms: standard of care combined with ERY001
Drug: Gemcitabine
Drug: 5-fluoro-uracil/oxaliplatin/leucovorin (folfox) — oxaliplatin 85 mg/m2 levo-leucovorin 200 mg/m2 5-FU 400 mg/m2

SUMMARY:
A new approach that aims to destroy pancreatic tumor cells through modification of the tumor environment.

Asparagine synthetase (ASNS) is an enzyme wich synthetise asparagine. Asparagine is an essential nutriment for pancreatic cancer cells which have no or low level of ASNS.

by L-asparaginase encapsulated in erythrocytes deplete (supress) Plasma asparagine.

in selected patients having no or low ASNS, may provide a new therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

A patient is eligible for the study if all of the following criteria are met:

* Advanced or metastatic exocrine pancreatic adenocarcinoma, confirmed histologically
* Available archival tumor tissue block with sufficient tissue either from primary tumor and/or from metastatic lesions for biomarker testing; alternatively, unstained slides with sufficient tissue may be substituted
* Only 1 prior systemic therapy for advanced or metastatic disease. NOTE: Patient must be eligible to 2nd line gemcitabine or mFOLFOX6 treatment Documented disease progression during or following first-line therapy for advanced disease
* Measurable lesion (>1cm) as assessed by CT scan or MRI (Magnetic Resonance Imaging) according to RECIST criteria (version 1.1)
* Age 18 years and older
* ECOG performance status 0 or 1
* Ability to understand, and willingness to sign, a written informed consent and to comply with the scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Patient beneficiary of a Social Security Insurance if applicable

Exclusion Criteria:

A patient is excluded from the study if any of the following criteria are met:

* Patient who have received Oxaliplatin in first line will not be eligible in FOLFOX arm; Patient who received Gemcitabine in first line will not be eligible in Gemcitabine arm
* Resectable pancreatic adenocarcinoma
* Known hypersensitivity to L-asparaginase or have had prior exposure to any form of L-asparaginase
* Anti-vitamin K treatment. Replacement with low molecular weight heparin treatment if required
* Inadequate organ functions:

  * hemoglobin < 9.0 g/dl, neutrophil count < 1.5 x 109/L, platelets < 100 x 109/L.
  * Liver or pancreatic function abnormalities

    * AST or ALT > 3 x ULN, or
    * Total bilirubin > 1.5 x ULN, or
    * Lipase > 2 x ULN with suggestive clinical sign of pancreatitis or > 3N without suggestive clinical sign
  * Renal insufficiency: Renal clearance determined by the Cockroft and Gault Formula < 60 mL/min
* Current or prior coagulopathy disorders in the last month

  * PT ≥1.5 fold the upper limit of normal value or
  * INR ≥1.5 fold the upper limit of normal value or
  * Fibrinogen ≤ 0.75 fold the lower limit of normal value
* Known Infection: HIV, active hepatitis related to B or C virus
* Concurrent active malignancies (with the exception of in situ carcinoma of the cervix and inactive non melanoma skin cancer
* Other serious conditions than pancreatic cancer according to investigator's opinion
* NYHA Grade ≥ 2 congestive heart failure
* Systemic chemotherapy or radiation within the last 3 weeks or major surgery within 4 weeks NOTE: chemotherapy or radiation therapy given in less than 3 weeks is allowed, provided patient recovered from all related toxicities
* History of grade 3 blood transfusion reaction (life threatening situation)
* Presence of anti-erythrocyte antibodies (auto-antibodies or anti-public antibodies) preventing from getting a compatible packed Red Blood Cells for the patient
* Participation in another concurrent clinical trial
* Women of child-bearing potential and men with partners of childbearing potential without effective contraception as well as pregnant or breast feeding women
* Other severe acute/chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From last study treatment assessment visit until patient's death, loss to follow up, or study closure, assessed up to 36 months.
  Evaluate the effects of eryaspase when combined with chemotherapy for the second line treatment of patients with pancreatic adenocarcinoma in terms of OS, whose tumors has low or no ASNS expression (ASNS 0 or 1+)
Progression free survival (PFS) | From date of randomization to first documented progression of disease, death for any cause or until start of new anti-cancer treatment, whcihever came first, assessed up to 24 months.
  Evaluate the effects of eryaspase when combined with chemotherapy for the second line treatment of patients with pancreatic adenocarcinoma in terms of PFS, whose tumors has low or no ASNS expression (ASNS 0 or 1+)

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (Safety and Tolerability) | collected from time of informed consent until 4 weeks after last study treatment
  Compare the safety profile in patients treated with eryaspase in combination with chemotherapy versus chemotherapy alone, including adverse events, vital signs and clinical laboratory assessments
Overall survival | From last study treatment assessment visit until patient's death, loss to follow up, or study closure, assessed up to 36 months.
  Evaluate the effects of eryaspase in combination with chemotherapy on investigator-assessed OS in all randomized patients (all patients) and in patients with ASNS 2+/3+ expressing tumors.
Progression free survival | From date of randomization to first documented progression of disease, death for any cause or until start of new anti-cancer treatment, whcihever came first, assessed up to 24 months.
  Evaluate the effects of eryaspase in combination with chemotherapy on investigator-assessed PFS in all randomized patients (all patients) and in patients with ASNS 2+/3+ expressing tumors.
Objective response rate (ORR) | From date of randomization to last tumor assessment data collected for each patient, assessed up to 24 months.
  Evaluate the effect of eryaspase in combination with chemotherapy on the ORR, and the duration in all comers, patients with ASNS 0/1+ expressing tumors, and those with ASNS 2+/3+ expressing tumors.
Disease control rate (DCR) | From date of randomization to 16 and 24 weeks.
  Evaluate the effect of eryaspase in combination with chemotherapy on the DCR in all comers, patients with ASNS 0/1+ expressing tumors, and those with ASNS 2+/3+ expressing tumors.
Duration of response (DoR) | From date of first response of complete or partial response until tumor progression, assessed up to 24 months.
  Evaluate the effect of eryaspase in combination with chemotherapy on the DoR in all comers, patients with ASNS 0/1+ expressing tumors, and those with ASNS 2+/3+ expressing tumors.
Evaluate the relationship of clinical outcomes with tumor markers | From date of randomiztion to end of treatment visit, assessed up to 20 months.
  Evaluate the relationship of clinical outcome (i.e. OS, PFS, ORR, DCR and DoR) with tumor markers, namely cancer antigen (CA19-9), and carcinoembryonic antigen test (CEA).
Optical density reading | From date of randomization to first documented progression of disease, death for any cause or until start of new anti-cancer treatment, whcihever came first, assessed up to 24 months.
  Assess the effect of eryaspase in combination with chemotherapy on PFS, OS, ORR, BOR, and other clinical outcomes in ASNS subsets, as determined by optical density reading.
Quality of Life status | From date of randomiztion to end of treatment visit, assessed up to 20 months.
  Compare the 2 treatment arms with respect to change in quality of life status, the change of QOL relative to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Hammel, Pr MD, Principal Investigator — Hopital Beaujon
Locations (16):
- France (16):
  - Saint Catherine Institute, Avignon
  - Institut de Cancerologie, Brest
  - Hopital Beaujon, Clichy
  - Hospital Henri Mondor, Créteil
  - Groupe Hospitalier Mutualiste Grenoble, Grenoble
  - Centre Hospitalier Departemental Vendee - Les Oudairies, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Cnetre Leon Berard, Lyon
  - Institut Regional du Cancer-Montpellier Val d'Aurelle, Montpellier
  - Institute Mutualiste Montsouris, Paris
  - Hospital Saint Antoine, Paris
  - Hospital Pitie Salpetriere, Paris
  - CHU de Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Toulouse - Rangueil, Toulouse
  - CHU de Tours, Tours

REFERENCES:
- [Derived] Bachet JB, Blons H, Hammel P, Hariry IE, Portales F, Mineur L, Metges JP, Mulot C, Bourreau C, Cain J, Cros J, Laurent-Puig P. Circulating Tumor DNA is Prognostic and Potentially Predictive of Eryaspase Efficacy in Second-line in Patients with Advanced Pancreatic Adenocarcinoma. Clin Cancer Res. 2020 Oct 1;26(19):5208-5216. doi: 10.1158/1078-0432.CCR-20-0950. Epub 2020 Jun 30. PMID 32605910
- [Derived] Hammel P, Fabienne P, Mineur L, Metges JP, Andre T, De La Fouchardiere C, Louvet C, El Hajbi F, Faroux R, Guimbaud R, Tougeron D, Bouche O, Lecomte T, Rebischung C, Tournigand C, Cros J, Kay R, Hamm A, Gupta A, Bachet JB, El Hariry I. Erythrocyte-encapsulated asparaginase (eryaspase) combined with chemotherapy in second-line treatment of advanced pancreatic cancer: An open-label, randomized Phase IIb trial. Eur J Cancer. 2020 Jan;124:91-101. doi: 10.1016/j.ejca.2019.10.020. Epub 2019 Nov 21. PMID 31760314